CLINICAL TRIAL: NCT05324345
Title: The Construction and Application of a Web-based Home Multimodal Prehabilitation Program in Patients Undergoing Thoracic and Major Abdominal Surgeries: a Single-arm Clinical Trial
Brief Title: Web-based Home Multimodal Prehabilitation for Patients Undergoing Major Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LZJ004
Record Dates: First submitted 2022-03-31; First posted 2022-04-12 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Perioperative Recovery, Prehabilitation
Keywords: Internet medicine, Prehabilitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prehabilitation group (Experimental): This is a prospective single-arm study. All patients enrolled in this study will receive the multimodal prehabilitation strategy by the network learning platform after a complete assessment.
  Interventions: Behavioral: Prehabilitation group

INTERVENTIONS:
Behavioral: Prehabilitation group — All patients will be guided to use the network learning platform which including details in text, pictures and videos of their individualized prehabilitation strategy after a complete assessment. Multimodal prehabilitation strategy includes conventional guidance (including preoperative anesthesia assessment, drug treatment recommendations for chronic disease, quit smoking and abstinence), physical exercise (moderate aerobic exercise combined with resistance exercise and respiratory training), nutritional suggestion and optimization (whey protein supplement), and psychological therapy. All movements can be practiced with the reference to the standard videos in the network learning platform. Patients will check the prehabilitation content daily and form their own training tasks in the network learning platform. Standardized short message interviews will be sent to patients twice a week to optimize adherence and promote timely feedback.

SUMMARY:
Prehabilitation is the process of optimizing physical functionality preoperatively to enable the individual to maintain a normal level of function during and after surgery. Prehabilitation training based on aerobic exercise, resistance exercise, breathing exercise, nutrition supplement and physiology management preoperatively could have a positive effect on the recovery of postoperative functional capacity in patients undergoing surgery.

Investigators try to construct a short home-based multimodal prehabilitation model based on internetwork in order to improve the efficiency of prehabilitation training, enhance the compliance of patients, and reduce the medical human resources and economic burden. In this study, prehabilitation guidance would be given to preoperative patients through network learning platform. Short-term multi-modal family strategy intervention would perform during the preoperative waiting period, and patients could upload their training records and obtain personalized training guidance by network learning platform follow-up management mode. Investigators would evaluate the feasibility of this model and evaluate its impact on improving the perioperative functional status and prognosis of patients.

DETAILED DESCRIPTION:
Trimodal or multimodal prehabilitation strategy including exercise, diet and psychologic guidance could improve postoperative functional recovery for patients undergoing surgery. The development of internet medical provides possibility to improve the efficiency of patients' preoperative education, enhance the accuracy of prehabilitation execution, and reduce the medical human resources and economic burden.

This study tries to build the patient-centered network education and follow-up management based on the internet learning platform.

This is a prospective arm study. A total of 40 patients scheduled to have elective major thoracic, abdominal and retroperitoneal surgery (including thoracoscopic and laparoscopic surgery) will be recruited in this research at Peking Union Medical College Hospital. After informed consent is obtained, the baseline data (including basic information, past medical history, initial 6-minute walk distance, grip strength, pulmonary function et.al) will be collected. All patients will be guided to use the network learning platform which including details in text, pictures and videos of their individualized prehabilitation strategy after a complete assessment. Prehabilitation strategy is as follows: (1) quit smoking and abstinence; (2) a 5-minute warm-up exercise and a 25-minute aerobic exercise in the form of power walking, jogging, or cycling at least 3 times a week; (3) anaerobic exercise in form of bodyweight muscle training or pull strap training at least twice a week; (4) patients scheduled to have elective thoracic surgery also need to do breathing exercise in the form of blowing balloons, blowing the respiratory exerciser Tri-Ball, and active cycle of breathing techniques at least twice a day, 10 minutes each time; (5) nutritional advice and whey protein supplement 1 hour prior to exercise (20g/day for male and 15g/day for female patients); (6) psychological therapy by listening to soothing music and other relaxing activities. All details can be practiced with the reference to the standard videos in thenetwork learning platform. Patients will check the prehabilitation content daily and form their own training tasks in the network learning platform. Standardized short message interviews will be sent to patients twice a week to optimize adherence and promote timely feedback.

The length of prehabilitation will be 2-3 weeks, determined by the waiting time till surgery alone. After admission, the utilization rate of the prehabilitation network learning platform, the implementation of the prehabilitation strategy and the satisfaction with the network learning platform will be collected. Change of the following indicators from baseline to 1 day before surgery will be collected. The primary outcome is the change in 6-minute walk distance (6MWD), measured as functional walking capacity. The secondary outcomes include body-mass index(BMI), smoking cessation rate, grip strength, forced expiratory volume in 1 s (FEV1), forced vital capacity (FVC), FEV1/FVC, Duke Activity Status Index(DASI), Nutritional risk screening scale (NRS-2002), and Hospital Anxiety and Depression Scale (HADS).

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients in Peking Union Medical College Hospital between May 2022 to December 2022
2. From 18y/o to 70y/o
3. Decide to take the elective thoracic surgery or major abdominal surgery (including retroperitoneal surgery) in Peking Union Medical College Hospital.

Exclusion Criteria:

1. Decline to participant the study (due to any reason)
2. American Society of Anesthesiologists (ASA) grade >III
3. Patients plan to receive neoadjuvant therapy
4. Unable to cooperate (including mental disorder, conscious disturbance, and dysgnosia)
5. Unable to tolerate prehabilitation or aerobic strategy (including exercise guide, whey protein and psycho-relaxation exercise)
6. Unable to use a smartphone or unable to read Chinese
7. Local anesthesia or low-risk surgery (superficial surgery, outpatient surgery, or anticipated operation time <1 hour);
8. People who have an average of more than 90 minutes of moderate intensity aerobic exercise or more than 60 minutes of high intensity exercise per week.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in 6-minute walk distance | baseline, 1 day before surgery
  Use the change in 6-minute walk distance (6MWD) to evaluate the impact of prehabilitation on functional capability before surgery.

SECONDARY OUTCOMES:
Body mass index (BMI) | baseline, 1 day before surgery
  Body mass index (BMI) will be calculated by formula: BMI=weight(kg)/height(m)^2.
Smoking cessation rate | baseline, 1 day before surgery
  The number of smokers will be collected at baseline and 1 day before surgery, and smoking cessation rates will be calculated.
Grip strength | baseline, 1 day before surgery
  The grip strength of the hand will be measured by a grip strength tester (Jamar Plus+ Hand Evaluation Kit).
Forced expiratory volume in 1 s(FEV1) | baseline, 1 day before surgery
  Forced expiratory volume in 1 s (FEV1) of pulmonary function will be measured in liters.
Forced vital capacity (FVC) | baseline, 1 day before surgery
  Forced vital capacity (FVC) of pulmonary function will be measured in liters.
Forced expiratory volume in 1 s / Forced vital capacity (FEV1/FVC) | baseline, 1 day before surgery
  FEV1/FVC will be calculated with the FEV1 and FVC value and reported in percentage.
Duke Activity Status Index (DASI) | baseline, 1 day before surgery
  Evaluate the patients'functional capacity. The Duke Activity Status Index (DASI) is a 12-item scale (in the form of a self-administered questionnaire) that correlates well with peak oxygen uptake (Spearman correlation coefficient 0.80). DASI score is calculated by adding the points of all performed activities together. The higher the score (ranges from 0 to 58.2) the higher the functional status.
Nutritional risk screening scale (NRS-2002) | baseline, 1 day before surgery
  Evaluate the patients' nutritional risk. NRS includes assessment of the patient's disease severity (stress metabolism due to the degree of disease) and nutritional status (based on weight loss, body mass index (BMI) and general condition or food intake). Each section is scored from 0 to 3 points, and patients receive an extra point if they are 70 years or older.
Hospital Anxiety and Depression Scale (HADS) | baseline, 1 day before surgery
  The HADS is a questionnaire composed of 14 questions to screen for anxiety and depression. The questionnaire features 7 questions on anxiety and seven on depression. The maximum score for either anxiety or depression is 21 and the minimum for either is 0. The severity of anxiety and depression correlates with the scoring. HADS will be used to evaluate the impact of prehabilitation of mental capability.

CONTACTS AND LOCATIONS:
Overall Officials: Zijia LIU, M.D., Study Chair — Peking Union Medical College Hospital, Chinese Academy of Medicine Sciences